CLINICAL TRIAL: NCT01666418
Title: Pilot Study Investigating the Metabolic Activity and Transcriptional Profiling in Vivo in Tumor Biopsies in Melanoma Patients During Treatment With Pazopanib Alone and in Combination With Paclitaxel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZ10ON01
Record Dates: First submitted 2012-08-08; First posted 2012-08-16 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — pazopanib; Paclitaxel

ARMS (1):
- Pazopanib/Paclitaxel (Other)
  Interventions: Drug: Pazopanib/Paclitaxel

INTERVENTIONS:
Drug: Pazopanib/Paclitaxel

SUMMARY:
This is an open, monocentric, pilot study to determine the metabolic activity (glucose-uptake) in vivo during monotherapy with pazopanib in comparison to combination therapy with pazopanib plus paclitaxel and to investigate the transcriptional profile of cutaneous melanoma metastasis before and during the therapy (pazopanib vs. pazopanib plus paclitaxel) in subjects with unresectable Stage III or Stage IV melanoma who have not received prior cytotoxic chemotherapy.

Primary Objective:

Evaluation of metabolic activity in vivo

Secondary Objective:

Determination of changes in gene expression profiling Evaluation of the antitumor activity of the combination in terms of progression free survival (PFS). Changes in S100 and LDH during therapy at the same time points as FDG-PET/CT (a combined serum measurement of S100 and LDH)

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* Diagnosis of histologically or cytologically confirmed melanoma stage III or IV.
* Fresh tumor tissue must be provided for all subjects for biomarker analysis before (within 14 days prior to treatment start) and during (on day 10 of the pazopanib monotherapy and the last day of the treatment with pazopanib, day 70) treatment with investigational product (asservation in RNAlater, for kryo asservation, and for cell cultures)
* Assessable metastases (skin or superficial lymph nodes with a minimal diameter 1 cm)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ system function

Exclusion criteria:

* Prior malignancy.
* Central nervous system (CNS) metastases
* Corrected QT interval (QTc) > 480 msecs using Bazett's formula.
* History of any one or more of the following cardiovascular conditions within the past 6 months:

  * Cardiac angioplasty or stenting;
  * Myocardial infarction;
  * Unstable angina;
  * Coronary artery bypass graft surgery;
  * Symptomatic peripheral vascular disease;
  * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA).
* Poorly controlled hypertension
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
* Presence of uncontrolled infection
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding
* Evidence of active bleeding or bleeding diathesis
* Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity, except alopecia.
* Prior exposure to the study drug pazopanib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-08; Primary Completion 2014-10 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of metabolic activity in vivo | 84 days ( Baseline, Day 10, Day 70)
  The primary efficacy objective is to evaluate the metabolic activity in vivo through standardising the uptake value (SUV) in the FDG-PET/CT in comparison of the SUV between baseline, after pazopanib alone (day 10) and after pazopanib plus paclitaxel (day 70).

SECONDARY OUTCOMES:
Determination of changes in gene expression profiling | 84 days ( Baseline, Day 10, Day 70)
  Determination of changes in gene expression profiling on exon level in all patients with (sub)-cutaneous or superficial lymph node metastases (of melanoma) during pazopanib and pazopanib plus paclitaxel therapy in comparison to pretreatment profile
Evaluation of the antitumor activity of the combination in terms of progression free survival (PFS) | 112 days
Changes in S100 and LDH during therapy at the same time points as FDG-PET/CT (a combined serum measurement of S100 and LDH) | 84 days ( Baseline, Day 10, Day 70)

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Dummer, Professor MD, Principal Investigator — University Hospital Zurich, Division of Dermatology
Locations (1):
- University Hospital Zurich, Division of Dermatology, Zurich, Switzerland